CLINICAL TRIAL: NCT05326178
Title: Evaluating the Efficacy and the Acceptability of the Website "Ich Bin Alles" to Improve Depression Literacy in Parents of Healthy Adolescents Without a Mental Health Condition
Brief Title: Evaluation of a Website to Improve Depression Literacy in Parents of Healthy Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Prof. Otto Beisheim Foundation (Other)
Responsible Party: Principal Investigator, Ellen Greimel, Working group leader, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20116_2
Record Dates: First submitted 2022-04-01; First posted 2022-04-13 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Depressive Disorder; Depression in Adolescence
Keywords: Knowledge; Mental Health; Depression Literacy; Website; Online; Adolescence; Youth; Parental Behaviour
MeSH Terms: conditions — Depressive Disorder; Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- General information about depression (Experimental): Exposure to general information about depression
  Interventions: Other: General information about depression

INTERVENTIONS:
Other: General information about depression — Before starting the intervention, the participants are told that they will be shown parts of a website about depression. The participants are instructed to carefully attend to the website (e.g., to read the text precisely, to hear attentively to the podcasts and to view carefully the videos and images on the website). The time window spent for the reception of each part of the website are fixed.
  The participants will be shown parts of the website regarding general information about depression.

SUMMARY:
The aim of this study is to evaluate the efficacy and acceptability of the website "ich bin alles" (https://www.ich-bin-alles.de/) to improve depression literacy (knowledge about depression, which aid the recognition, treatment or prevention of depression) in parents of healthy adolescents without a mental health condition. The investigators will examine whether the website improves depression literacy in parents of adolescents aged 12 to 18 years without a mental health condition. The investigators will also assess the acceptability of the website among the participants.

DETAILED DESCRIPTION:
Few young people with major depressive disorder seek professional treatment in time. Concerns about social stigma, confidentiality, and limited knowledge about mental health conditions, such as depression, or mental health services are some of the main barriers to seek treatment. Increasing parents' knowledge about and attitude towards depression and mental health in childhood and adolescence is important to sensitize parents and increase their awareness towards depression and mental health in their children. These aspects might play a crucial role for parents to support their children's mental health, notice potential depressive symptoms in their children, react appropriately and take action if necessary. To address these issues and to contribute to knowledge gain in this target group, we developed an evidence-based website "ich bin alles" with two separate sub-websites for (1) adolescents (https://www.ich-bin-alles.de/) and (2) parents (…../eltern) to improve depression literacy in these groups.

To improve depression literacy in parents, the website provides general information for parents about depression in childhood and adolescence (e.g., symptoms, causes, course and treatment of depression). Furthermore, the website provides information about strategies for parents on how to support their children if they are affected by depression and on appropriate prevention strategies; i.e., strategies for promoting mental health (e.g., providing a healthy environment, reducing stress, undertaking positive activities, positive parenting), which are meant to serve as an addition to professional treatments of depression or to promote mental health in adolescents.

Target groups of the website are parents of adolescents aged 12 to 18 years with a history of depression, as well as parents of healthy adolescents aged 12 to 18 years. Easy access to information about depression would make early recognition of depression more likely and engage parents to help their children to seek help for depression.

Since the website targets two different groups, the investigators will evaluate the website accordingly:

Target group 1: Parents of adolescents with a major depressive disorder (acute or remitted) Target group 2: Parents of healthy adolescents (without a mental health condition)

The current study will focus on target group 2. A study focusing on target group 1 can be found in a separately registered clinical trial on clinicaltrials.gov.

The primary aim of this study is to evaluate the efficacy and acceptability of the website "ich bin alles" (https://www.ich-bin-alles.de/) to improve depression literacy in parents of healthy adolescents without a mental health condition.

ELIGIBILITY:
Inclusion Criteria:

* The absence of a current or remitted diagnosis of any psychiatric disorder in the participants' children is assessed using a semi-structured clinical interview: the "Kinder-DIPS". The Kinder-DIPS is a well-established German interview for the diagnosis of a wide range of axis I psychiatric disorders in children from ages six to 18.

Exclusion Criteria:

* Insufficient knowledge of German

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Change in Depression Literacy - Depression in children and adolescents as psychiatric disorder | Pre-Test, Post-Test (within 2 hours), Follow-Up (Week 4)
  This self-designed questionnaire is a self-report inventory to assess knowledge of depression in children and adolescents (frequency and comorbidities, treatment, symptoms, causes and course of depression; 26 items), with higher scores indicating more knowledge of depression as psychiatric disorder. Participants will complete this self-designed questionnaire at pre-test, post-test and follow-up to determine change in knowledge of depression in children and adolescents.

SECONDARY OUTCOMES:
Visual Aesthetics of Websites Inventory Short Version (VisAWI-S) | Post-Test (within 2 hours)
  The short version of the Visual Aesthetics of Websites Inventory (VisAWI-S) is self-report inventory to assess the evaluation of the website's design - especially the perceived visual aesthetics. Participants indicate their response to the four items (e.g., "The layout appears professionally designed") on a seven-point Likert scale (ranging from 1 "do not agree at all" to 7 "do fully agree").
Overall reception of the website | Post-Test (within 2 hours)
  The overall reception of the website as measured with a self-designed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Schulte-Körne, Professor, Study Director — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University Hospital Munich
Locations (1):
- Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University Hospital Munich, Munich, Germany, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Data in our study contains sensitive participant information, such as sociodemographic information. Since participants could possibly be identified by making our raw data publicly available, ethical principles of protecting participant confidentiality would be breached. Aggregated group data can be made available upon request.